CLINICAL TRIAL: NCT02261961
Title: Immune Function and Muscle Adaptations to Resistance Exercise in Older Adults
Acronym: TDAP2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: E1203-R; RX001203 (Other Grant/Funding Number: VA Rehabilitation R&D Application); 608119 (Other: CAVHS Institutional Review Board)
Record Dates: First submitted 2014-09-19; First posted 2014-10-10 (Estimated); Results first posted 2021-09-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-08

CONDITIONS: Sarcopenia; Aging; Immune Function
Keywords: resistance exercise; Juven; exercise training; interleukin-1; insulin-like growth factor
MeSH Terms: conditions — Sarcopenia | interventions — Tetanus Toxoid; Resistance Training; Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nutritional Supplement (Experimental): Subjects in the supplement group will consume orange-flavored Muscle Armor according to the manufacturer's directions: one serving (approximately 30g, i.e. one scoop provided with the product by its manufacturer), twice daily mixed with 12 ounces (oz) of water beginning after all baseline assessments are performed including assessment of the response to acute exercise and continuing until the end of study participation.
  Interventions: Biological: TDAP; Other: Acute Resistance Exercise; Other: Resistance Exercise Training; Other: Post-training Follow-up; Dietary Supplement: Nutritional Supplement (Muscle Armor)
- Placebo (Placebo Comparator): Subjects in the placebo group will consume orange-flavored Kool-Aid (Kraft Foods) according to the manufacturer's directions: one serving (approximately 13g, i.e. one scoop provided with the product by the pharmacy), twice daily mixed with 12 ounces (oz) of water beginning after all baseline assessments are performed including assessment of the response to acute exercise and continuing until the end of study participation.
  Interventions: Biological: TDAP; Other: Acute Resistance Exercise; Other: Resistance Exercise Training; Other: Post-training Follow-up; Dietary Supplement: Placebo (Kool-Aid)

INTERVENTIONS:
Biological: TDAP — Both arms will receive the tetanus, diptheria, and pertussis vaccination after two weeks of treatment with supplement or placebo
  Other Names: tetanus, diptheria, and pertussis vaccination
Other: Acute Resistance Exercise — Both arms will receive a single bout of resistance exercise twice, before and after two weeks of treatment with supplement or placebo, and be evaluated for the response within blood and muscle
  Other Names: Single bout of exercise
Other: Resistance Exercise Training — Both arms will receive 36 sessions of progressive high-intensity resistance exercise training (thigh muscle) over the course of approximately 12 weeks.
  Other Names: Chronic exercise
Other: Post-training Follow-up — Both arms will continue to receive treatment with supplement or placebo for approximately 26 weeks after completion of the exercise training. During this time subjects will not be allowed to perform resistance exercise.
  Other Names: Detraining Period
Dietary Supplement: Nutritional Supplement (Muscle Armor) — Subjects in the supplement group will consume orange-flavored Muscle Armor according to the manufacturer's directions: one serving (approximately 30g, i.e. one scoop provided with the product by its manufacturer), twice daily mixed with 12 ounces (oz) of water beginning after all baseline assessments are performed including assessment of the response to acute exercise and continuing until the end of study participation.
  Arms: Nutritional Supplement
Dietary Supplement: Placebo (Kool-Aid) — Subjects in the placebo group will consume orange-flavored Kool-Aid (Kraft Foods) according to the manufacturer's directions: one serving (approximately 13g, i.e. one scoop provided with the product by the pharmacy), twice daily mixed with 12 ounces (oz) of water beginning after all baseline assessments are performed including assessment of the response to acute exercise and continuing until the end of study participation.
  Arms: Placebo

SUMMARY:
The loss of muscle mass and strength due to aging leads to serious health problems for older adults. Muscle health can be improved by exercise training, but some people improve their strength substantially, whereas others improve little. The reason for this variation is unknown. This study will investigate whether function of the immune system influences how well people respond to exercise. Older Veterans who participate will have their muscle size, strength, and function measured periodically for almost a year. Participants will drink a nutritional supplement or placebo daily and complete a 36 session strength training program. Participants will be vaccinated for tetanus and donate small amounts of blood and muscle tissue during the study so that immune function can be compared to muscle outcomes during training and during a long-term follow-up. The study results should increase the investigators' understanding of the negative effects of aging on muscle and will possibly lead to better strategies for muscle maintenance and rehabilitation for older adults.

DETAILED DESCRIPTION:
Objective: The study will examine the influence of immune function in older adults on improvement of muscle mass, strength, and function by resistance training. The maintenance of those benefits during long term follow-up will also be examined. This objective will be accomplished by a double-blind randomized placebo-controlled trial of a nutritional supplement (Muscle Armor) which evidence suggests can improve immune function, promote muscle growth, and counteract muscle loss. The study premise is that aging results in decreased ability of the immune system to respond to stimuli such as exercise. The study proposes that the supplement will improve muscle health by promoting a shift in immune function of older adults from a pro-inflammatory state towards a state which supports muscle growth and maintenance.

Research Plan: The study will randomize Veterans (age 60-80, N=50) to participate in the supplement or placebo groups in a three phase study. The phases of participation correspond to the three specific aims. Aim 1 will determine if 2-weeks of supplementation improves immune function. Humoral immune function will be assessed as the response to vaccination. Innate immune function will be measured as systemic and cellular responses to acute resistance exercise that the investigators' previous studies indicate are affected by aging. Aim 2 will determine if supplementation during 36 sessions of progressive high-intensity resistance training boosts improvement in muscle size (CT scan), strength, and function (gait and balance). Muscle adaptations at the cellular levels will also be measured. Aim 3 will determine if continued supplementation for 26-weeks after completion of exercise training promotes the retention of the gains in muscle size, strength, and function. Multivariable testing will then be used to compare the results between Aims 1, 2, and 3 to determine whether or not immune function is correlated with muscle adaptation to training or detraining.

Methods: Participants will undergo nine blood draws and five muscle biopsies of the vastus lateralis over the course of the study so that the effects of the supplement on immune function and cellular adaptations to training can be measured. Three of the blood draws will be used to assess the antibody response to the tetanus, pertussis, and diphtheria vaccine. Muscle and blood will be collected before and after a bout of exercise conducted before and after the 2-weeks of supplementation prior to training. Immune function will be measured using the blood based on pro- and anti-inflammatory cytokine levels, the balance between specific T-cell subpopulations, and the proliferative capacity of mononuclear cells. Immune function will be measured in muscle based on macrophage content of specific cytokines and growth factors. The investigators' previous study showed that these muscle measures strongly correlate with size and strength gain after training. Key signaling pathways including nuclear factor-k B and PI3 kinase will also be measured. The fifth biopsy will be collected post-training to measure adaptation at the cellular level based on changes in number of satellite cells and myonuclei and fiber size. Hypotheses related to these measures will be tested with 80% power to detect at least 0.8 standard deviations difference in means between the supplement and placebo groups.

Clinical Relevance: Exercise is clearly able to affect immune function. However, the proposed study will attempt to modulate immune function and determine the effects on exercise outcomes. The study will also examine detraining, an important issue for older adults, that is usually omitted from training studies. Thus, the study will potentially advance the understanding of the mechanisms of muscle gain and loss in older adults, but more importantly, the study will evaluate a nutritional intervention as a complement to exercise for supporting muscle health during aging. Targeting the immune system may be the advantage needed for an older Veteran to successfully maintain or restore the muscle mass, strength, and function that is necessary for personal independence.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* Age 60-80 years
* Body Mass Index of 18.5 - 29.9 kg/m2

Exclusion Criteria:

* Currently participating in any other research study involving an intervention
* Smokes tobacco products
* Tetanus or TDAP vaccine in previous two years
* Allergic to vaccination
* Seizure in past 3 months
* Guillain-Barre Syndrome in past 3 months
* Takes the medications heparin, plavix / clopidogrel, or coumadin / warfarin
* Allergic to lidocaine
* Significant problem with fainting
* Problems walking or exercising with both legs
* Participated in a weight-lifting program targeting the thighs in last 3 months
* Pains, tightness or pressure in chest during physical activity
* Metastatic cancer or undergoing chemotherapy
* Cerebral aneurysm or intracranial bleed in past year
* End-stage congestive heart failure (NYHA Stage IV)
* Unstable abdominal or thoracic aortic aneurysm (>4cm)
* Renal disease requiring dialysis
* Allergic to vaccination
* Acute retinal hemorrhage or ophthalmologic surgery in past 3 months
* Bone fractures in the pelvis, legs, or feet in the last 3 months
* Hernia that causes pain during physical activity
* Myocardial infarction or cardiac surgery in past 3 months
* Pulmonary embolism or deep venous thrombosis in past 3 months
* Proliferative diabetic retinopathy or severe nonproliferative retinopathy
* Active suicidality or suicidal ideation
* Systemic bacterial infection
* Taking aspirin in any form and unable/unwilling to discontinue at least 10 days prior to muscle biopsy
* Unwilling to halt concurrent use of amino acid or protein supplements
* Unwilling to halt new use of nutritional supplements
* Unwilling to maintain current normal diet
* Encephalopathy in past 7 days
* Active oral or genital herpes
* Current use of appetite stimulants
* Current treatment for mania or bipolar disorder or taking lithium.
* Diagnosis of a significant cognitive deficit
* Untreated severe aortic stenosis
* Uncontrolled diabetes mellitus (HbA1C>10)
* Uncontrolled hypertension or hypotension (>160/100, <100 systolic)
* Uncontrolled malignant cardiac arrhythmia
* Unstable angina
* Allergic to latex or tape
* Bleeding or clotting disorders
* Taking any non-ASA NSAID and unable or unwilling to discontinue use for 3 days prior to muscle biopsy
* Taking Fish Oil, Gingko, Garlic, Saw Palmetto, Turmeric, or Vitamin E and unable or unwilling to discontinue use for 10 days prior to the muscle biopsy procedure
* Significant problems with chronic pain
* Uncontrolled asthma or allergies
* Taking lactulose, nitrates plus hypertension medications or Viagra
* Liver cirrhosis or other severe liver disease
* History of peripheral artery disease
* Certain Steroid or androgen use in past 3 months
* Other physician judgment
* Significantly abnormal complete blood count (CBC) or prothrombin time (PT)/partial thromboplastin time (PTT)/international normalized ratio (INR)

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2014-07-23 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Dennis, PhD, Principal Investigator — Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR
Locations (1):
- Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR, North Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Long DE, Villasante Tezanos AG, Wise JN, Kern PA, Bamman MM, Peterson CA, Dennis RA. A guide for using NIH Image J for single slice cross-sectional area and composition analysis of the thigh from computed tomography. PLoS One. 2019 Feb 7;14(2):e0211629. doi: 10.1371/journal.pone.0211629. eCollection 2019. PMID 30730923
- [Result] Dennis RA, Long DE, Landes RD, Padala KP, Padala PR, Garner KK, Wise JN, Peterson CA, Sullivan DH. Tutorial for using SliceOmatic to calculate thigh area and composition from computed tomography images from older adults. PLoS One. 2018 Oct 2;13(10):e0204529. doi: 10.1371/journal.pone.0204529. eCollection 2018. PMID 30278056
- [Result] Kosmac K, Peck BD, Walton RG, Mula J, Kern PA, Bamman MM, Dennis RA, Jacobs CA, Lattermann C, Johnson DL, Peterson CA. Immunohistochemical Identification of Human Skeletal Muscle Macrophages. Bio Protoc. 2018 Jun 20;8(12):e2883. doi: 10.21769/BioProtoc.2883. PMID 30148186
- [Result] Dennis RA, Ponnappan U, Kodell RL, Garner KK, Parkes CM, Bopp MM, Padala KP, Peterson CA, Padala PR, Sullivan DH. Immune Function and Muscle Adaptations to Resistance exercise in Older Adults: Study Protocol for a Randomized Controlled Trial of a Nutritional Supplement. Trials. 2015 Mar 27;16:121. doi: 10.1186/s13063-015-0631-3. PMID 25872570

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 59 consented but only 44 randomized due to 15 either being excluded or withdrawal prior to randomization
Groups:
- Nutritional Supplement: Subjects in the supplement group will consume orange-flavored Muscle Armor according to the manufacturer's directions: one serving (approximately 30g, i.e. one scoop provided with the product by its manufacturer), twice daily mixed with 12 ounces (oz) of water beginning after all baseline assessments are performed including assessment of the response to acute exercise and continuing until the end of study participation.
  TDAP: Both arms will receive the tetanus, diptheria, and pertussis vaccination after two weeks of treatment with supplement or placebo
  Acute Resistance Exercise: Both arms will receive a single bout of resistance exercise twice, before and after two weeks of treatment with supplement or placebo, and be evaluated for the response within blood and muscle
  Resistance Exercise Training: Both arms will receive 36 sessions of progressive high-intensity resistance exercise training (thigh muscle) over the course of approx 12 weeks.
Period: Overall Study
Arm/Group | Nutritional Supplement | Placebo
Started | 22 | 22
Completed | 13 | 20 (One subject listed as completed who withdrew but finished training phase and has usable data.)
Not Completed | 9 | 2

BASELINE CHARACTERISTICS:
Population: Included subjects who completed all or majority of study
Groups:
- Nutritional Supplement: Subjects in the supplement group will consume orange-flavored Muscle Armor according to the manufacturer's directions: one serving (approximately 30g, i.e. one scoop provided with the product by its manufacturer), twice daily mixed with 12 ounces (oz) of water beginning after all baseline assessments are performed including assessment of the response to acute exercise and continuing until the end of study participation.
  TDAP: Both arms will receive the tetanus, diptheria, and pertussis vaccination after two weeks of treatment with supplement or placebo
  Acute Resistance Exercise: Both arms will receive a single bout of resistance exercise twice, before and after two weeks of treatment with supplement or placebo, and be evaluated for the response within blood and muscle
  Resistance Exercise Training: Both arms will receive 36 sessions of progressive high-intensity resistance exercise training (thigh muscle) over the course of approx 12 wks and undergo a post-training Follow-up
- Placebo: Subjects in the placebo group will consume orange-flavored Kool-Aid (Kraft Foods) according to the manufacturer's directions: one serving (approx 13g, i.e. one scoop provided with the product by the pharmacy), twice daily mixed with 12 ounces (oz) of water beginning after all baseline assessments are performed including assessment of the response to acute exercise and continuing until the end of study participation.
  TDAP: Both arms will receive the tetanus, diptheria, and pertussis vaccination after two weeks of treatment with supplement or placebo
  Acute Resistance Exercise: Both arms will receive a single bout of resistance exercise twice, before and after two weeks of treatment with supplement or placebo, and be evaluated for the response within blood and muscle
  Resistance Exercise Training: Both arms will receive 36 sessions of progressive high-intensity resistance exercise training (thigh muscle) over the course of approx 12 wks and undergo a Post-training Follow-up
- Total: Total of all reporting groups
Arm/Group | Nutritional Supplement | Placebo | Total
Number analyzed (Participants) | 13 | 20 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 4 | 6
  >=65 years | 11 | 16 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] — Age measured in years
  years | 69.3 (4.8) | 69.1 (5.0) | 69.2 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 12 | 19 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 9 | 15 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 20 | 33
Leg Press [Mean (Standard Deviation); unit: pounds] — strength in one-repetition max
  pounds | 486.7 (112.1) | 519.3 (130.6) | 499.5 (118.8)
Knee Curl [Mean (Standard Deviation); unit: pounds] — strength in one-repetition max
  pounds | 135.7 (37.1) | 128.2 (26.5) | 130.9 (30.7)
Knee Extension [Mean (Standard Deviation); unit: pounds] — strength in one-repetition max
  pounds | 136.7 (37.1) | 132.3 (37.9) | 134.0 (37.1)
Muscle Size [Mean (Standard Deviation); unit: centimeters squared] — cross sectional area of thigh
  centimeters squared | 144.5 (22.2) | 139.1 (21.0) | 141.2 (21.3)
Tetanus Antibody Levels [Mean (Standard Deviation); unit: units per ml] — ELISA measure of blood antibody levels to antigen
  units per ml | 4.3 (2.1) | 3.7 (2.5) | 3.9 (2.3)
Pertussis Antibody Levels [Mean (Standard Deviation); unit: units per ml] — ELISA measure of blood antibody levels to antigen
  units per ml | 48.8 (32.9) | 59.7 (41.2) | 55.4 (38.0)
Diptheria Antibody Levels [Mean (Standard Deviation); unit: units per ml] — ELISA measure of blood antibody levels to antigen
  units per ml | 0.6 (0.7) | 0.7 (1.0) | 0.7 (0.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Plasma Concentration of Antibodies to Pertussis Antigen (1 Week Post-vaccine)
Description: The change in plasma antibody concentration for response to the pertussis antigen within the tetanus, diphtheria, and pertussis (TDAP) vaccination will be measured between baseline and one week post-vaccination.
Time Frame: change from baseline at 1 week post-vaccine
Measure: Mean (Standard Deviation); unit: units per ml
Groups:
- Nutritional Supplement: Subjects in the supplement group will consume Muscle Armor according to the manufacturer's directions: one serving (approximately 30g, i.e. one scoop provided with the product by its manufacturer), twice daily mixed with 12 ounces (oz) of water beginning after all baseline assessments including assessment of the response to acute exercise and continuing until the end of study participation.
  TDAP: Both arms will receive the tetanus, diptheria, and pertussis vaccination after two weeks of treatment with supplement or placebo
  Acute Resistance Exercise: Both arms will receive a single bout of resistance exercise twice, before and after two weeks of treatment with supplement or placebo, and be evaluated for the response within blood and muscle
  Resistance Exercise Training: Both arms will receive 36 sessions of progressive high-intensity resistance exercise training (thigh muscle) over the course of approximately 12 weeks.
  Post-training Follow-up: B
- Placebo: Subjects in the placebo group will consume orange-flavored Kool-Aid (Kraft Foods) according to the manufacturer's directions: one serving (approximately 13g, i.e. one scoop provided with the product by the pharmacy), twice daily mixed with 12 ounces (oz) of water beginning after all baseline assessments including assessment of the response to acute exercise and continuing until the end of study participation.
  TDAP: Both arms will receive the tetanus, diptheria, and pertussis vaccination after two weeks of treatment with supplement or placebo
  Acute Resistance Exercise: Both arms will receive a single bout of resistance exercise twice, before and after two weeks of treatment with supplement or placebo, and be evaluated for the response within blood and muscle
  Resistance Exercise Training: Both arms will receive 36 sessions of progressive high-intensity resistance exercise training (thigh muscle) over the course of approximately 12 weeks.
  Post-training Follow-up
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 13 | 20
units per ml | 63.1 (39.7) | 63.2 (40.7)
Statistical Analysis 1: Comparison: Nutritional Supplement vs Placebo; Test type: Superiority; p > 0.05, ANCOVA; Slope = -0.24275

2. Primary Outcome: Change in Plasma Concentration of Antibodies to Pertussis Antigen (2 Weeks Post-vaccine)
Description: The change in plasma antibody concentration for response to the pertussis antigen within the tetanus, diphtheria, and pertussis (TDAP) vaccination will be measured between baseline and two weeks post-vaccination.
Time Frame: change from baseline at 2 weeks post-vaccine
Measure: Mean (Standard Deviation); unit: units per ml
Groups:
- Nutritional Supplement: Subjects in the supplement group will consume orange-flavored Muscle Armor according to the manufacturer's directions: one serving (approximately 30g, i.e. one scoop provided with the product by its manufacturer), twice daily mixed with 12 ounces (oz) of water beginning after all baseline assessments including assessment of the response to acute exercise and continuing until the end of study participation.
  TDAP: Both arms will receive the tetanus, diptheria, and pertussis vaccination after two weeks of treatment with supplement or placebo
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 13 | 20
units per ml | 159.2 (130.7) | 216.7 (240.1)
Statistical Analysis 1: Comparison: Nutritional Supplement vs Placebo; Test type: Superiority; p > 0.05, ANCOVA; Slope = 1.3707

3. Primary Outcome: Change in Plasma Concentration of C-Reactive Protein
Description: Plasma c-reactive protein will be measured before and after two weeks of treatment with supplement or placebo.
Time Frame: change from baseline at 2 weeks of treatment
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 13 | 20
mg/L | 0.34 (1.52) | -3.96 (10.05)

4. Primary Outcome: Change in the Number of Muscle Macrophages Per Myofiber (Pre- to Post-acute Exercise)
Description: The change in the number of muscle macrophages per myofiber will be calculated for muscle collected before and 72 hours after a single bout of resistance exercise. The changes in macrophage numbers before and after two weeks of treatment with supplement or placebo will be compared.
Time Frame: change from baseline at 2 weeks of treatment
Population: The overall number of participants analyzed was less than the total number of participants due to insufficient specimen.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 9 | 10
percent change | 16.01 (49.36) | -8.54 (25.70)

5. Primary Outcome: Change in Muscle Strength After Exercise Training for 12 Weeks
Description: The change in muscle strength after exercise training will be measured as the difference in one-repetition maximum capability for knee extension from before and after completion of the exercise training program.
Time Frame: change from baseline at completion of exercise training phase (12 weeks)
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 13 | 20
pounds | 195.4 (54.4) | 182.9 (45.7)
Statistical Analysis 1: Comparison: Nutritional Supplement vs Placebo; Test type: Superiority; p > 0.05, ANCOVA; Slope = -0.35579

6. Secondary Outcome: Change in Plasma Concentration of Antibodies to Tetanus Antigen (1 Week Post-vaccine)
Description: The change in plasma antibody concentration for response to the tetanus antigen within the tetanus, diphtheria, and pertussis (TDAP) vaccination will be measured between baseline and one week post-vaccination.
Time Frame: change from baseline at 1 week post-vaccine
Measure: Mean (Standard Deviation); unit: units per ml
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 13 | 20
units per ml | 5.6 (2.4) | 4.1 (2.6)
Statistical Analysis 1: Comparison: Nutritional Supplement vs Placebo; Test type: Superiority; p > 0.05, ANCOVA; Slope = 0.004493

7. Secondary Outcome: Change in Plasma Concentration of Antibodies to Tetanus Antigen (2 Weeks Post-vaccine)
Description: The change in plasma antibody concentration for response to the tetanus antigen within the tetanus, diphtheria, and pertussis (TDAP) vaccination will be measured between baseline and two weeks post-vaccination.
Time Frame: change from baseline at 2 weeks post-vaccine
Measure: Mean (Standard Deviation); unit: units per ml
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 13 | 20
units per ml | 8.6 (3.7) | 8.2 (5.1)
Statistical Analysis 1: Comparison: Nutritional Supplement vs Placebo; Test type: Superiority; p > 0.05, ANCOVA; Slope = 0.870653

8. Secondary Outcome: Change in Plasma Concentration of Antibodies to Diptheria Antigen (1 Week Post-vaccine)
Description: The change in plasma antibody concentration for response to the diptheria antigen within the tetanus, diphtheria, and pertussis (TDAP) vaccination will be measured between baseline and one week post-vaccination.
Time Frame: change from baseline at 1 week post-vaccine
Measure: Mean (Standard Deviation); unit: units per ml
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 13 | 20
units per ml | 1.1 (1.2) | 1.1 (1.4)
Statistical Analysis 1: Comparison: Nutritional Supplement vs Placebo; Test type: Superiority; p > 0.05, ANCOVA; Slope = -0.38664

9. Secondary Outcome: Change in Plasma Concentration of Antibodies to Diptheria Antigen (2 Weeks Post-vaccine)
Description: The change in plasma antibody concentration for response to the diptheria antigen within the tetanus, diphtheria, and pertussis (TDAP) vaccination will be measured between baseline and two weeks post-vaccination.
Time Frame: change from baseline at 2 weeks post-vaccine
Measure: Mean (Standard Deviation); unit: units per ml
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 13 | 20
units per ml | 2.1 (1.6) | 1.7 (1.5)
Statistical Analysis 1: Comparison: Nutritional Supplement vs Placebo; Outcomes were compared as percent change from the baseline measure using multiple methods by a blinded statistician. Differences between groups were assessed using ANCOVA, Welch's t-test, and Wilcoxon. No significant differences were found between groups for any outcome regardless of method used; Test type: Superiority; p > 0.05, ANCOVA; Slope = 0.335124

10. Secondary Outcome: Number of Muscle Macrophages Per Myofiber (Resting)
Description: The number of muscle macrophages per myofiber will be counted for resting muscle collected before and after two weeks of treatment with supplement or placebo.
Time Frame: change from baseline at 2 weeks of treatment
Population: The overall number of participants analyzed was less than the total number of participants due to insufficient specimen.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 9 | 10
percent change | 6.89 (21.99) | 42.42 (51.74)

11. Secondary Outcome: Change in Muscle Size After Exercise Training for 12 Weeks
Description: The change in size of the thigh muscle group after exercise training will be measured as the difference in cross-sectional area based on CT scan before and after completion of the exercise training program.
Time Frame: change from baseline at completion of exercise training phase (12 weeks)
Measure: Mean (Standard Deviation); unit: centimeters squared
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 13 | 20
centimeters squared | 155.8 (24.1) | 146.4 (22.6)
Statistical Analysis 1: Comparison: Nutritional Supplement vs Placebo; Test type: Superiority; p > 0.05, ANCOVA; Slope = 0.03145

12. Secondary Outcome: Change in Muscle Strength at Week 16 of the Post-Training Period
Description: The change in muscle strength (one-repetition maximum for knee extension) after completion of the exercise training program will be measured during a follow-up period lacking exercise.
Time Frame: difference between baseline and time point one of de-training follow-up period (week 16)
Population: The overall number of participants analyzed was less than the total number of participants due to a participant not completing entire study.
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 13 | 19
pounds | 175.5 (50.0) | 162.9 (34.5)
Statistical Analysis 1: Comparison: Nutritional Supplement vs Placebo; Test type: Superiority; p > 0.05, ANCOVA; Slope = -0.43902

13. Secondary Outcome: Change in Balance After Exercise Training for 12 Weeks
Description: The change in balance ability after exercise training will be measured as the difference in Berg Balance Scale (Min 0, Max 56, Higher is Better) score between before and after completion of the exercise training program.
Time Frame: change from baseline at completion of exercise training (12 weeks)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 13 | 19
score on a scale | 0.54 (1.27) | 0.79 (1.23)

14. Secondary Outcome: Change in Balance During the Post-Training Period at 26 Weeks of the Post-training Period
Description: The change in balance based on the Berg Balance Scale (Min 0, Max 56, Higher is Better) score will be measured during a follow-up period lacking exercise after completion of the exercise training program.
Time Frame: difference between time of training completion and time point two of de-training follow-up period (26 weeks)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 13 | 19
score on a scale | 0.08 (0.49) | 0.05 (1.27)

15. Secondary Outcome: Change in Balance at Week 16 of the Post-Training Period
Description: as for outcome 14
Time Frame: difference between time of training completion and time point one of de-training follow-up period (week 16)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 13 | 19
score on a scale | -0.08 (0.49) | 0.11 (0.32)

16. Secondary Outcome: Change in Walking Ability After Exercise Training for 12 Weeks
Description: The change in walking ability after exercise training will be measured using the six minute walk test, i.e. the distance the participant can walk without shortness of breath in six minutes.
Time Frame: change from baseline at completion of exercise training (12 weeks)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 13 | 19
meters | 18.03 (31.74) | 22.25 (40.91)

17. Secondary Outcome: Change in Walking Ability at Week 16 of the Post-Training Period
Description: The change in walking ability based on the six-minute walk test will be measured during a follow-up period lacking exercise after completion of the exercise training program.
Time Frame: difference between end of training and time point one of de-training follow-up period (week 16)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 13 | 19
meters | -13.62 (38.91) | -29.02 (55.89)

18. Secondary Outcome: Change in Walking Ability at Week 26 of the Post-Training Period
Description: as for outcome 17
Time Frame: difference between end of training and time point two of de-training follow-up period (week 26)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 13 | 19
meters | 1.34 (38.24) | -20.85 (52.33)

19. Secondary Outcome: Change in Gait Speed After Exercise Training for 12 Weeks
Description: The change in gait speed ability after exercise training will be measured as the difference in habitual walking speed for 10 meters before and after completion of the exercise training program.
Time Frame: change from baseline at completion of exercise training (12 weeks)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 13 | 19
meters per second | 0.04 (0.11) | 0.05 (0.14)

20. Secondary Outcome: Change in Gait Speed at Week 16 of the Post-Training Period
Description: The change in habitual walking speed over 10 meters will be measured as the difference between values at the end of the training program and time points during a follow-up period lacking exercise.
Time Frame: difference between after training and time point one of de-training follow-up period (week 16)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 13 | 19
meters per second | -0.02 (0.10) | -0.03 (0.14)

21. Secondary Outcome: Change in Gait Speed During at Week 26 of the Post-Training Period
Description: as for outcome 20
Time Frame: difference between after training and time point two of de-training follow-up period (week 26)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 13 | 19
meters per second | 0.04 (0.13) | 0.03 (0.14)

22. Secondary Outcome: Change in Muscle Size at Week 26 of the Post-Training Period
Description: The change in size of the thigh muscle group during the post-training period will be measured as the difference in cross-sectional area based on CT scan at the end of the training program and at the end of study participation.
Time Frame: difference between baseline and time point two of de-training follow-up period (week 26)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: centimeters squared
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 13 | 19
centimeters squared | 143.6 (24.4) | 140.5 (19.9)
Statistical Analysis 1: Comparison: Nutritional Supplement vs Placebo; Test type: Superiority; p > 0.05, ANCOVA; Slope = -0.07603

23. Secondary Outcome: Change in Timed Up and Go After Exercise Training for 12 Weeks
Description: The change in time required to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down will be measured as the difference between before and after completion of the exercise training program.
Time Frame: change from baseline at completion of exercise training (12 weeks)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 13 | 19
seconds | -0.22 (0.65) | -0.26 (0.71)

24. Secondary Outcome: Change in Timed Up and Go at Week 16 of the Post-Training Period
Description: The change in time required to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down will be measured as the difference between time points at the end of the training program and during the post-training period.
Time Frame: difference between after training and time point one of de-training follow-up period (week 16)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 13 | 19
seconds | 0.33 (1.12) | 0.18 (0.77)

25. Secondary Outcome: Change in Timed Up and Go at Week 26 of the Post-Training Period
Description: as for outcome 24
Time Frame: difference between after training and time point two of de-training follow-up period (week 26)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 13 | 19
seconds | 0.14 (1.18) | -0.15 (0.65)

26. Secondary Outcome: Percent Change in Resting Muscle Concentration of Interleukin-1 Beta
Description: The muscle concentration of interleukin-1 beta will be measured before and after two weeks of treatment with supplement or placebo.
Time Frame: change from baseline at 2 weeks of treatment
Population: The overall number of participants analyzed was less than the total number of participants due to insufficient specimen.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 7 | 7
percent change | 58.00 (172.57) | 40.93 (148.80)

27. Secondary Outcome: Change in Muscle Concentration of Interleukin-1 Beta (Pre- to Post-acute Exercise)
Description: The change in the muscle concentration of interleukin-1 beta before and one hour after a single bout of resistance exercise. The changes in macrophage numbers before and after two weeks of treatment with supplement or placebo will be compared.
Time Frame: change from baseline at 2 weeks of treatment
Population: The overall number of participants analyzed was less than the total number of participants due to insufficient specimen.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 7 | 7
percent change | 110.52 (424.92) | -89.70 (2744.35)

28. Secondary Outcome: Change in Resting Muscle Atrophy Gene MURF Expression
Description: The change in resting muscle atrophy gene MURF expression will be measured before and after two weeks of treatment with supplement or placebo.
Time Frame: percent change from baseline at 2 weeks of treatment
Population: The overall number of participants analyzed was less than the total number of participants due to insufficient specimen.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 12 | 18
percent change | 20.98 (99.61) | 148.17 (325.87)

29. Secondary Outcome: Change in Resting Muscle Atrophy Gene MURF Expression (Post-acute Exercise)
Description: The change in resting muscle atrophy gene MURF expression will be measured before and 72 hours after a single bout of exercise completed before and after two weeks of treatment with supplement or placebo.
Time Frame: change from baseline at 2 weeks of treatment
Population: The overall number of participants analyzed was less than the total number of participants due to insufficient specimen.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 12 | 17
percent change | 38.69 (224.53) | -76.98 (423.64)

30. Secondary Outcome: Change in Resting Muscle Protein Kinase B
Description: The change in resting muscle Protein Kinase B will be measured before and after two weeks of treatment with supplement or placebo.
Time Frame: change from baseline at 2 weeks of treatment
Population: The overall number of participants analyzed was less than the total number of participants due to insufficient specimen.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 9 | 9
percent change | 78.15 (187.21) | 51.24 (112.35)

31. Secondary Outcome: Change in Muscle Protein Kinase B (Post-acute Exercise)
Description: The change in muscle Protein Kinase B will be measured before and 72 hours after a single bout of exercise completed before and after two weeks of treatment with supplement or placebo.
Time Frame: change from baseline at 2 weeks of treatment
Population: The overall number of participants analyzed was less than the total number of participants due to insufficient specimen.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 9 | 9
percent change | -27.24 (127.78) | 9.48 (85.32)

32. Secondary Outcome: Change in Number of Muscle Satellite Cells After Exercise Training for 12 Weeks
Description: The change in the satellite cell content of muscle will be measured as the difference in the number of satellite cells in muscle before and after completion of the exercise training program.
Time Frame: change from baseline at completion of exercise training (12 weeks)
Population: The overall number of participants analyzed was less than the total number of participants due to insufficient specimen.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 12 | 16
percent change | 18.24 (48.93) | 9.96 (40.72)

33. Secondary Outcome: Change in Number of Myonuclei After Exercise Training for 12 Weeks
Description: The change in the myonuclear content of muscle will be measured as the difference in the number of myonuclei in muscle before and after completion of the exercise training program.
Time Frame: change from baseline at completion of exercise training (12 weeks)
Population: The overall number of participants analyzed was less than the total number of participants due to insufficient specimen.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 12 | 16
percent change | 6.88 (36.99) | 20.28 (27.65)

34. Secondary Outcome: Change in Muscle Fiber Size After Exercise Training for 12 Weeks
Description: The change in the muscle fiber size will be measured as the difference in fiber size before and after completion of the exercise training program.
Time Frame: change from baseline at completion of exercise training (12 weeks)
Population: The overall number of participants analyzed was less than the total number of participants due to insufficient specimen.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 10 | 15
percent change | 35.26 (51.59) | 47.28 (54.87)

35. Other Pre Specified Outcome: Plasma Concentration of Aspartate Aminotransferase After Product Consumption for 15 Weeks
Description: Plasma aspartate aminotransferase will be measured as a safety indicator of liver function at baseline, after completion of the exercise training program, and at the end of the study.
Time Frame: at completion of the exercise training program (15 weeks)
Population: The overall number of participants analyzed was less than the total number of participants due to a clinical lab error and a participant not completing entire study.
Measure: Mean (Standard Deviation); unit: Units/L
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 12 | 19
Units/L | 29.25 (7.79) | 26.37 (7.78)

36. Other Pre Specified Outcome: Plasma Concentration of Alanine Aminotransferase After Product Consumption for 15 Weeks
Description: Plasma Alanine Aminotransferase will be measured as a safety indicator of liver function at baseline, after completion of the exercise training program, and at the end of the study.
Time Frame: completion of the exercise training program (15 weeks)
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: Units/L
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 12 | 19
Units/L | 24.83 (13.90) | 24.53 (13.21)

37. Other Pre Specified Outcome: Ratio of Plasma Concentrations of Blood Urea Nitrogen to Creatinine After Product Consumption for 15 Weeks
Description: Plasma blood urea nitrogen and creatinine will be measured as a safety indicator of kidney function at baseline, after completion of the exercise training program, and at the end of the study.
Time Frame: completion of the exercise training program (15 weeks)
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 12 | 19
ratio | 20.40 (5.22) | 13.35 (3.98)

38. Other Pre Specified Outcome: Plasma Concentration of Aspartate Aminotransferase After 42 Weeks of Product Consumption
Description: as for outcome 35
Time Frame: end of study (42 weeks)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units/L
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 13 | 19
Units/L | 28.31 (8.83) | 27.16 (9.50)

39. Other Pre Specified Outcome: Plasma Concentration of Alanine Aminotransferase After 42 Weeks of Product Consumption
Description: as for outcome 36
Time Frame: end of study (42 weeks)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units/L
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 13 | 19
Units/L | 22.38 (8.49) | 25.32 (10.11)

40. Other Pre Specified Outcome: Ratio of Plasma Concentrations of Blood Urea Nitrogen to Creatinine After 42 Weeks of Product Consumption
Description: as for outcome 37
Time Frame: end of study (42 weeks)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 13 | 19
ratio | 20.98 (9.10) | 14.44 (4.95)

41. Other Pre Specified Outcome: Change in Muscle Strength at Week 26 of the Post-Training Period
Description: as for outcome 12
Time Frame: difference between baseline and time point two of de-training follow-up period (week 26)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 13 | 19
pounds | 171.2 (50.6) | 165.0 (36.3)
Statistical Analysis 1: Comparison: Nutritional Supplement vs Placebo; Test type: Superiority; p > 0.05, ANCOVA; Slope = -0.4745

42. Other Pre Specified Outcome: Plasma Concentration of Aspartate Aminotransferase
Description: as for outcome 35
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: Units/L
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 13 | 20
Units/L | 26.62 (7.52) | 27.55 (10.97)

43. Other Pre Specified Outcome: Plasma Concentration of Alanine Aminotransferase
Description: as for outcome 36
Time Frame: baseline
Population: The overall number of participants analyzed was less than the total number of participants due to clinical lab error.
Measure: Mean (Standard Deviation); unit: Units/L
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 13 | 19
Units/L | 21.54 (6.24) | 27.42 (16.68)

44. Other Pre Specified Outcome: Ratio of Plasma Concentrations of Blood Urea Nitrogen to Creatinine
Description: as for outcome 37
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Nutritional Supplement | Placebo
Number analyzed (Participants) | 13 | 20
ratio | 14.06 (3.75) | 14.52 (5.18)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from participants at every interaction (in-person, phone contact, or monitoring of electronic health record prior to in-person appointment) from the point of informed consent until 30 days after participant completion of study, which averaged 62 weeks total.
Groups:
- Nutritional Supplement: Subjects in the supplement group will consume orange-flavored Muscle Armor according to the manufacturer's directions beginning after all baseline assessments are performed including assessment of the response to acute exercise and continuing until the end of study participation.
  TDAP: Both arms will receive the tetanus, diptheria, and pertussis vaccination after two weeks of treatment with supplement or placebo
  Acute Resistance Exercise: Both arms will receive a single bout of resistance exercise twice, before and after two weeks of treatment with supplement or placebo, and be evaluated for the response within blood and muscle
  Resistance Exercise Training: Both arms will receive 36 sessions of progressive high-intensity resistance exercise training (thigh muscle) over the course of approximately 12 weeks.
  Post-training Follow-up: Both arms will continue to receive treatment with supplement or placebo for approximately 26 weeks after completion of the exercise training.
- Placebo: Subjects in the placebo group will consume orange-flavored Kool-Aid (Kraft Foods) according to the manufacturer's directions beginning after all baseline assessments are performed including assessment of the response to acute exercise and continuing until the end of study participation.
  TDAP: Both arms will receive the tetanus, diptheria, and pertussis vaccination after two weeks of treatment with supplement or placebo
  Acute Resistance Exercise: Both arms will receive a single bout of resistance exercise twice, before and after two weeks of treatment with supplement or placebo, and be evaluated for the response within blood and muscle
  Resistance Exercise Training: Both arms will receive 36 sessions of progressive high-intensity resistance exercise training (thigh muscle) over the course of approximately 12 weeks.
  Post-training Follow-up: Both arms will continue to receive treatment with supplement or placebo for approx 26 wks after completion of the ex training.
Arm/Group | Nutritional Supplement | Placebo
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 4/22 | 7/22
Other Adverse Events (participants affected / at risk) | 11/22 | 16/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nutritional Supplement (N=22) | Placebo (N=22)
SAE (Cardiac disorders) | 0 (0) | 0 (0) — Prior to randomization one subject withdrew for unstated health reasons and one was excluded due to chest pain.
cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cardiovascular Event (Cardiac disorders) | 1 (1) | 2 (2)
colon polyps (Gastrointestinal disorders) | 1 (1) | 0 (0)
gallstones (Hepatobiliary disorders) | 0 (0) | 2 (2)
lost name and address (Product Issues) | 2 (2) | 3 (3)
knee surgery (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
unknown surgery (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nutritional Supplement (N=22) | Placebo (N=22)
biopsy pain or bruise (General disorders) | 2 (2) | 3 (3)
bodily wound (General disorders) | 1 (1) | 3 (3)
cold, flu, or infection (General disorders) | 3 (3) | 5 (5)
gastrointestinal distress (Gastrointestinal disorders) | 1 (1) | 3 (3)
musculoskeletal soreness, strain, or pain (Musculoskeletal and connective tissue disorders) | 4 (7) | 7 (11)
skin irritation, rash, or numbness (Skin and subcutaneous tissue disorders) | 3 (3) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-06-26): https://cdn.clinicaltrials.gov/large-docs/61/NCT02261961/Prot_SAP_000.pdf
  • Informed Consent Form (2016-05-11): https://cdn.clinicaltrials.gov/large-docs/61/NCT02261961/ICF_001.pdf